CLINICAL TRIAL: NCT06236126
Title: Prospective, Single-Center, Randomized, Double-Blind, Clinical Trial for The Evaluation of Pain Associated to The Epidural Tuohy Needle Insertion With Prior Administration of Subcutaneous or Intradermal Lidocaine in Parturient Women Requesting Epidural Analgesia for Laboring Pain.
Brief Title: SKIN WHEAL - Subcutaneous or Intradermal Lidocaine in Epidural for Laboring Pain.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ling-Qun Hu, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023H0250
Record Dates: First submitted 2024-01-12; First posted 2024-02-01 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Analgesia, Obstetrical
MeSH Terms: conditions — Agnosia | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: A single center, prospective, randomized, double blind pilot study for the evaluation of pain due to epidural Tuohy needle insertion with prior administration of subcutaneous or intradermal administration of lidocaine in parturient women requesting epidural analgesia for laboring pain at The Ohio State University Wexner Medical Center - Obstetric Anesthesia Division.
Who Masked: Participant, Outcomes Assessor
Masking Description: A blinded observer (positioned in front of the patient and unable to see the procedure) will record data during the epidural procedure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTRADERMAL (Active Comparator): Prior to insertion of the Tuohy epidural needle, each patient will receive an injection of 3 mL 1% lidocaine either intradermally (Group Intradermal).
  Interventions: Procedure: 1% Lidocaine Injection
- SUBCUTANEOUS (Active Comparator): Prior to insertion of the Tuohy epidural needle, each patient will receive an injection of 3 mL 1% lidocaine subcutaneously (Group Subcutaneous).
  Interventions: Procedure: 1% Lidocaine Injection

INTERVENTIONS:
Procedure: 1% Lidocaine Injection — Prior to insertion of the Tuohy epidural needle, each patient will receive an injection of 3 mL 1% lidocaine either intradermally (Group Intradermal) or subcutaneously (Group Subcutaneous).

SUMMARY:
The purpose of this study is to explore the differences between the pain associated with epidural Tuohy needle insertion with prior administration of subcutaneous or intradermal lidocaine using two different pain assessment tools (numerical rate scale (NRS) and Critical-Care Pain Observation Tool (CPOT)) in parturient women requesting epidural analgesia for laboring pain. Subjects will go through the following study procedures: review of medical history prior to surgery. Subjects will be randomly assigned to one of the two study groups in a 1:1 ratio to one of the two different standard methods to administer lidocaine prior to epidural Tuohy needle insertion: intradermal or subcutaneous lidocaine administration. Prior to insertion of the Tuohy epidural needle, each patient will receive an injection of 3 mL 1% lidocaine either intradermally (Group Intradermal) or subcutaneously (Group Subcutaneous). A blinded observer (positioned in front of the patient and unable to see the procedure) will record baseline NRS scores, HR, and BP after the patient has been positioned for the epidural procedure and prior to the administration of lidocaine. During the procedure, the blinded observer will objectively record patient's vocal responses, facial expressions, bodily movements, and muscle tension (caused by pain reflex) using the CPOT and NRS scales during lidocaine administration and the first Tuohy needle insertion. After each injection, the blinded observer will record the corresponding heart rate. When the procedural anesthesiologist has exited the room, the blinded observer will then collect the patient's procedure satisfaction score from 0 (worst satisfaction) to 10 (most satisfaction) at the conclusion of the procedure. Likewise, the blinded observer will also collect the final post-procedure heart rate and blood pressure.

DETAILED DESCRIPTION:
EXPERIMENTAL METHODS Study design: A single center, prospective, randomized, double blind pilot study for the evaluation of pain due to epidural Tuohy needle insertion with prior administration of subcutaneous or intradermal administration of lidocaine in parturient women requesting epidural analgesia for laboring pain at The Ohio State University Wexner Medical Center - Obstetric Anesthesia Division.

Sample size: Since this is a pilot study, 25 patients with complete data in each group will be needed for the study, as no single study has been found to help sample size calculations. We estimated 25 patients per group (Intradermal Group and Subcutaneous Group) will be required to learn more about procedural pain on this patient population. However, we are requesting to consent 60 subjects in total, accounting for 20% of screen failure and/or early termination. A total of 60 patients will be included.

Study Population: Parturient women requesting epidural analgesia for laboring pain at The Ohio State University Wexner Medical Center - Obstetric Anesthesia Division.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Parturient women requesting epidural analgesia for laboring pain
* Ability to consent in English language

Exclusion Criteria:

* Women undergoing cesarean delivery.
* Administration of opioids in the 4 hours before study enrollment.
* Administration of IV magnesium sulfate within the last 24 hours.
* Diabetes mellitus (Type I and II).
* Neurocardiogenic signs or symptoms (e.g., dizziness, lightheadedness, bradycardia, and syncope) during IV cannulation.
* Cervical dilation >6 cm (if in labor).
* BMI ≥ 35.
* Spinal anesthesia.
* Chronic pain patients.
* Opioid use disorder
* Patient with intrauterine fetal demise
* Prisoners.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Parturient women requesting epidural analgesia for laboring pain at The Ohio State University Wexner Medical Center - Obstetric Anesthesia Division.
Enrollment: 50 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-11-13 (Estimated); Study Completion 2026-11-13 (Estimated)

PRIMARY OUTCOMES:
The Critical-Care Pain Observation Tool (CPOT) | Procedure (during lidocaine administration and at epidural Tuohy needle insertion)
  To assess the differences in The Critical-Care Pain Observation Tool pain scores (as units) during lidocaine administration and at epidural Tuohy needle insertion between both groups. The Critical-Care Pain Observation Tool (CPOT) includes four behavioral pain indicators (facial expressions, body movements, muscle tension and patient's vocalizations) to assess pain in critical care settings, rating pain levels with a score from 0-8.

SECONDARY OUTCOMES:
Numerical rating score (NRS) for pain | Procedure (during lidocaine administration and at epidural Tuohy needle insertion)
  To assess the differences in Numerical rating score (as units) pain scores during lidocaine administration (0, no pain; 10, worst pain imaginable) at epidural Tuohy needle insertion between both groups.
Blood pressure (BP) | at baseline, Procedure (during lidocaine administration and at epidural Tuohy needle insertion)
  To assess the differences in systolic and diastolic blood pressure (as mmHg) at baseline, lidocaine administration and epidural Tuohy needle insertion between both groups
Heart Rate (HR) | at baseline, Procedure (during lidocaine administration and at epidural Tuohy needle insertion)
  To • To assess the differences in heart rate (as beats per minute) at baseline, lidocaine administration and epidural Tuohy needle insertion between both groups
Patient procedural satisfaction score | at 30 minutes after the epidural procedure
  To assess the differences in overall patient procedural satisfaction score (0 indicated 'total discontent' and 10 'total satisfaction') between both groups

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
Fifty patients will be randomized into each group before the labor epidural procedure via a web-based REDCap by an unblinded research team member. Data collection forms will be used and recorded by a blinded research team member who will keep the data and add the data into the REDCap site. Both the study subjects and the research team members who collect data will be blinded.
  Results will be presented as mean ± SD or median with interquartile range. Normal distribution is assessed by descriptive statistics and histograms. Data are compared between groups by using student t-test, Chi-Square, or the Mann-Whitney U test accordingly. P < 0.05 is considered significant.